CLINICAL TRIAL: NCT00761540
Title: A Dose Escalation Study to Investigate the Pharmacokinetics, Tolerability and Safety of Liraglutide After Multiple s.c. Doses in Healthy Chinese Male Subjects
Brief Title: To Investigate the Blood Concentration of Liraglutide as Well as the Effects on Glucose and Insulin After 21 Days of Daily Subcutaneous Injections of Liraglutide or Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-3533
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- A1 (Experimental)
  Interventions: Drug: liraglutide
- A2 (Placebo Comparator)
  Interventions: Drug: placebo
- B1 (Experimental)
  Interventions: Drug: liraglutide
- B2 (Placebo Comparator)
  Interventions: Drug: placebo
- C1 (Experimental)
  Interventions: Drug: liraglutide
- C2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Liraglutide for s.c. injection once daily: dose step 1 (9 subjects)
  Arms: A1
Drug: placebo — Liraglutide placebo for s.c. injection once daily: dose step 1 (3 subjects)
  Arms: A2
Drug: liraglutide — Liraglutide for s.c. injection once daily: dose step 1, followed by dose step 2 (9 subjects)
  Arms: B1
Drug: placebo — Liraglutide placebo for s.c. injection once daily: dose step 1, followed by dose step 2 (3 subjects)
  Arms: B2
Drug: liraglutide — Liraglutide for s.c. injection once daily: dose step 1, followed by dose steps 2 and 3 (9 subjects)
  Arms: C1
Drug: placebo — Liraglutide placebo for s.c. injection once daily: dose step 1, followed by dose steps 2 and 3 (3 subjects)
  Arms: C2

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to investigate the blood concentration of liraglutide (pharmacokinetics) as well as the effects on glucose and insulin (pharmacodynamics) after 21 days of daily subcutaneous injections (injected under the skin) of liraglutide or placebo. In addition, the safety and tolerability of liraglutide will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial related activities
* Healthy Chinese male subjects
* Body mass index (BMI) between 19.0 and 27.0 kg/m2 (both inclusive)
* Fasting plasma glucose less than 6.0 mmol/L
* Non-smoker

Exclusion Criteria:

* Clinically significant abnormalities on pre-study clinical examination or any laboratory measurements during screening (any abnormality should be discussed with the clinical monitor)
* Presence of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders
* Blood pressure in supine position at the screening, after resting for 5 min, outside the ranges 90- 140 mmHg systolic and/or 40 - 90 mmHg diastolic
* Pulse in supine position at the screening, after resting for 5 min, outside the range 40 - 100 times/min
* Hepatitis B surface antigen, Hepatitis C antibodies or HIV antibodies positive.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
AUC 0-24h (last dosing day): Area under the plasma liraglutide curve from 0 to 24 hours after last dosing. | After 21 days of treatment

SECONDARY OUTCOMES:
AUC 0-24h: Area under the plasma liraglutide curve from 0 to 24 hours after first dosing, AUC0-24h (Day 1) | After 1 day of treatment
Adverse events | After 21 days of treatment
Hypoglycaemic events | After 21 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Jiang J, Zhang J, Jacobsen LV, Hu P. The pharmacokinetics, pharmacodynamics, and tolerability of liraglutide, a once-daily human GLP-1 analogue, after multiple subcutaneous administration in healthy Chinese male subjects. J Clin Pharmacol. 2011 Dec;51(12):1620-7. doi: 10.1177/0091270010389468. Epub 2011 Jan 27. PMID 21273395
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com